CLINICAL TRIAL: NCT03595605
Title: Association Between Inpatient Steps Per Day and Patient Functional Status/Disposition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-01792
Record Dates: First submitted 2018-05-22; First posted 2018-07-23 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Physical Medicine
MeSH Terms: interventions — Walking; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FitBit Group (Experimental): Will receive a wearable device (FitBit) designed to track number of steps for the duration of their hospital stay. They will receive nudges twice/day to ambulate
  Interventions: Behavioral: Ambulation
- Control Group-Standard of Care (Active Comparator): 300 subjects who will receive usual standard of care on a general inpatient medicine unit with the addition of a wearable device (FitBit) to track usual mobility in this setting. will complete their admission without push for increased activity (although having the device may influence their steps taken).
  Interventions: Other: Standard of Care

INTERVENTIONS:
Behavioral: Ambulation — This group will be encouraged twice daily to ambulate
  Arms: FitBit Group
Other: Standard of Care — Care as usual at inpatient NYU Langone
  Arms: Control Group-Standard of Care

SUMMARY:
This study will incorporate the use of wearable actigraphy devices (Fitbit) on research participants admitted to medicine inpatient units at Tisch Hospital and/or NYU Brooklyn. The investigator's sample size will be 600 randomized into two groups, with basic inclusion criteria including age greater than 65 years and pre-hospital ambulatory status. While both groups will be monitored in terms of their activity (specifically pedometer data), the intervention group will have twice daily encouragement of ambulation. Once a subject is enrolled, data will be collected daily and at time of discharge.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to acute inpatient medicine unit
* Ambulatory without assistive device prior to hospitalization
* Medical clearance to ambulate on the unit
* Active MyChart account or willing to activate MyChart account
* iOS or Android device

Exclusion Criteria:

* Patients less than or equal to 65 years old
* Not Admitted to acute inpatient medicine unit
* Ambulatory with assistive device prior to hospitalization
* No Medical clearance to ambulate on the unit
* Inactive MyChart account and not willing to activate MyChart account
* No iOS or Android device

In addition, an individual who meets any of the following criteria will be excluded from participation in this study:

* Oxygen requirement at rest
* Lower extremity prosthesis
* Admitted for joint replacement surgery
* History of frequent falls
* Admitted for syncope.
* If patients have specifically opted out of being contacted about research (visible in the Epic header while in their chart)
* Admitted from nursing home

Ages: 66 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Determine how many steps patients admitted to the medicine units are taking at baseline | 1 Day
  Steps will be measured using a wearable device (FitBit) designed to track number of steps for the duration of their hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Gavriil Ilizarov, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States